CLINICAL TRIAL: NCT04044014
Title: Prospective, Randomized Control Trial to Evaluate the Dermatological Reaction of Healthy Volunteers to Gellan Sheet and Fluid Gel Dressings (Gellan Contact Study)
Brief Title: Gellan Contact Study
Acronym: GCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Wellcome Trust (Other); University Hospital Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 189413
Record Dates: First submitted 2017-09-14; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2018-09

CONDITIONS: Thermal Injury; Skin Burn
Keywords: Gellan, thermal injury, healthy volunteers, skin
MeSH Terms: conditions — Paresthesia

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to receive the treatment dressing (either the Gellan sheet or Gellan fluid gel) on one arm (Left or Right), and the control dressing (Mepitel One) on the other arm. The first phase will be for 1 hour and the 2nd phase will be for 3 days.
Who Masked: Outcomes Assessor
Masking Description: Two assessors will be evaluating the skin for erythema, dryness and oedema. They will be blinded to which arm has received the treatment and control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A (Active Comparator): Left arm: Gellan sheet; Right arm: Mepitel One.
  Interventions: Device: Gellan sheet; Device: Mepitel One
- Arm B (Active Comparator): Left arm: Mepitel One; Right arm: Gellan sheet.
  Interventions: Device: Gellan sheet; Device: Mepitel One
- Arm C (Active Comparator): Left arm: Gellan fluid gel; Right arm: Mepitel One.
  Interventions: Device: Gellan fluid gel; Device: Mepitel One
- Arm D (Active Comparator): Left arm: Mepitel One; Right arm: Gellan fluid gel.
  Interventions: Device: Gellan fluid gel; Device: Mepitel One

INTERVENTIONS:
Device: Gellan sheet — Gellan sheet.
  Arms: Arm A; Arm B
Device: Gellan fluid gel — Gellan fluid gel.
  Arms: Arm C; Arm D
Device: Mepitel One — Control dressing-- Mepitel One.

SUMMARY:
The primary objective of this study will be to establish the safety of the two different Gellan formulations (sheet and fluid gel) following its application to the epidermis of healthy volunteers. This will be compared to a control dressing-- Mepitel One (Polyurethane net with soft Silicone).

DETAILED DESCRIPTION:
This contact study is part of the Wellcome trust Anti-scarring Dressing project to develop a carrier dressing that will be used to deliver therapeutic agents to the skin. A polysaccharide, Gellan, has been chosen as the main component of this dressing (the biomembrane)and it can be produced in either a sheet or fluid gel forms. Gellan is a widely used material in both the food and medical industry e.g. as a lubricant in eye-drops (e.g. Timoptol XE, Merck Sharp & Dohme, USA).

As part of the development of the dressing, the epidermal (skin) response to Gellan needs to be evaluated to check its safety.

The main objective of this study is to establish the safety of the two different Gellan formulations (2% Gellan sheet and 2% Gellan fluid gel) following application to the epidermis (skin).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥ 18 years old
* Subjects who can provide informed consent

Exclusion Criteria:

* Subject with existing skin conditions/diseases which may interfere with the aim(s) of the study. Examples include pathological fibrosis e.g. scleroderma; pathological thinning e.g. epidermolysis bullosa and collagen disorders e.g. Marfan's syndrome
* Chronic steroid use, history of skin malignancy or chronic papulo-squamous disease (e.g. eczema, pemphigus) and history of Steven Johnson or TENS disease
* Blemishes, marks (e.g. tattoos, scars or burns,) on the test site(s) which may interfere with assessment on the test site
* Use of medication which may affect may affect skin response
* Known allergy to the materials used in the study
* Known allergy to adhesive plasters or tapes
* Fitzpatrick skin type VI (due to the difficulty of identifying erythema)
* Irritated skin on the test site
* Known pregnancy (confirmed by urine pregnancy test) or lactating
* Inability to commit to attending all sessions.
* Participation in another study which may affect the results of this contact study.
* Any other reason that clinician considers will interfere with the objectives of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2017-02-13 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Skin reaction | 3 days (72 hours+/-3 hours)
  Skin will be evaluated for erythema, dryness and oedema by two observers using a visually based scale (Visual skin assessment scale; this is a novel scale devised by the research team).
  The scale is as follows:
  1. Erythema: 0-4 (Higher values are worse)
  2. Dryness: 0-3 (Higher values are worse)
  3. Oedema: 0-1 (Higher values are worse)
  Each subscale is evaluated individually and not combined.

SECONDARY OUTCOMES:
Participant satisfaction with dressing | At end of study (after 3 days)
  Participant satisfaction in terms of pain, itch, comfort and ease of removal (evaluated using a questionnaire).
  Name of questionnaire: "Participant evaluation questionnaire"
  Questions:
  1. Was the dressing comfortable? (Yes/No)
  2. Was there any itch? (Yes/No)
  3. Was there any pain? (Yes/No)
  4. Was the dressing comfortable to remove? (Yes/No)
Clinician satisfaction with dressing | At end of study (after 3 days)
  Clinician satisfaction in terms of ease of application, handling, removal, durability, conformity (evaluated using a questionnaire).
  Name of questionnaire: "Clinician evaluation questionnaire"
  Questions:
  1. Is the dressing still moist? (Yes/No)
  2. Is the dressing still intact? (Yes/No)
  3. Has any fragmentation occurred? (Yes/No)
  4. Has any tearing occurred? (Yes/No)

CONTACTS AND LOCATIONS:
Locations (1):
- Wellcome Trust Clinical Research Facility, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.